CLINICAL TRIAL: NCT00986947
Title: Phase 2 Study of IVIg and Rituximab for Desensitization of Highly Sensitized Deceased Donor Renal Transplantation Candidates
Brief Title: Desensitization of Highly Sensitized Deceased Donor Renal Transplantation Candidates
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00027111
Record Dates: First submitted 2009-09-29; First posted 2009-09-30 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Kidney Failure
MeSH Terms: conditions — Renal Insufficiency | interventions — Immunoglobulins, Intravenous; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IvIg with Rituximab (Experimental)
  Interventions: Drug: IVIg and rituximab

INTERVENTIONS:
Drug: IVIg and rituximab — A maximum of four doses (each single dose being 2gm/kg) of IVIg will be administered over a four-month period, with one dose administered each month. Each single dose of 2gm/kg will be administered in two half-doses (1gm/kg each) to be given one day apart, with one day of hemodialysis on the intervening day between the two half-doses.
  If a compatible kidney transplant organ offer is received, upon admission to the hospital and immediately prior to the transplant operation, patients will receive a single infusion of Rituximab (375 mg/m2 BSA).
  Other Names: Gamunex and Rituxan

SUMMARY:
Some patients who need kidney transplants have high levels of antibodies that make them incompatible with most potential deceased donor kidney offers. These patients are considered highly-sensitized and are very difficult to transplant because the likelihood that they will receive a compatible organ is very low. There are some medications and procedures that can decrease the antibody levels and this can increase the chance of finding a compatible donor for these patients. In this study the investigators will give two medications (IVIg and Rituximab) to highly-sensitized patients who are on the waiting list for a deceased donor kidney transplant. After the investigators administer these medications, the investigators will continue to check for compatibility as organ offers are received. If a compatible organ offer is received, the investigators will perform the transplant using that organ. The investigators hypothesize that these medications will lower antibody levels and increase the chance that a these patients are able to receive a compatible kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-75
* End-stage renal disease on dialysis
* Panel Reactive Antibody (PRA) > 60%
* Have been evaluated for and are currently listed for deceased donor renal transplantation

Exclusion Criteria:

* Have contraindication to transplantation
* Have contraindication to receiving IVIG
* Have allergy to IVIG
* Have received IVIG for desensitization previously without effect
* Pregnant women or those intending to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Medical Institutions, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 participants were enrolled.
Period: Overall Study
Arm/Group | IvIg With Rituximab
Started | 20
Completed | 0
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | IvIg With Rituximab
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Time to Kidney Transplantation
Time Frame: 4 months
Population: Data was not collected for this outcome measure. The study was terminated prematurely due to the P.I. leaving the institution.
Arm/Group | IvIg With Rituximab
Number analyzed (Participants) | 0

2. Secondary Outcome: Decrease in Panel Reactive Antibody
Time Frame: 4 months
Population: as for outcome 1
Arm/Group | IvIg With Rituximab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- IvIg With Rituximab: Intravenous immunoglobulin (IVIg) and rituximab: A maximum of four doses (each single dose being 2gm/kg) of IVIg will be administered over a four-month period, with one dose administered each month. Each single dose of 2gm/kg will be administered in two half-doses (1gm/kg each) to be given one day apart, with one day of hemodialysis on the intervening day between the two half-doses.
  If a compatible kidney transplant organ offer is received, upon admission to the hospital and immediately prior to the transplant operation, patients will receive a single infusion of Rituximab (375 mg/m2 BSA).
Arm/Group | IvIg With Rituximab
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes